CLINICAL TRIAL: NCT06212687
Title: Evaluation of a Digital Pre-therapy Patient Education Program (StartHjelp) in Outpatient Mental Health Care
Acronym: StartHjelp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 635362 b
Record Dates: First submitted 2023-12-01; First posted 2024-01-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Issue; Mental Disorder; Patient Education
Keywords: Patient education; Patient Satisfaction; Self Efficacy; Pre-therapy; DIgital health; Mental health; Therapy preparation
MeSH Terms: conditions — Mental Disorders; Patient Satisfaction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention is a pre-therapy informational app, presenting information about the treatment process, options, patient rights, user organizations, and self-help while on waiting list before mental health outpatient treatment. The information is delivered stepwise through video and text, while also providing links to additional information if needed. The videos are made available to the patients gradually, with more general information about the treatment process first, and more specific information as the first session approaches. The patient has the opportunity to rewatch the videos if needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital pre-therapy informational intervention (StartHjelp). (Experimental): Patients gets access to StartHjelp, an app which gradually present treatment relevant information while the patient is on waiting list for mental health outpatient services.
  Interventions: Behavioral: Digital pre-therapy patient education program (StartHjelp)
- Control group (Active Comparator): The control group gets sent all the same information as the intervention group in written form, by mail.
  Interventions: Behavioral: Comparator intervention

INTERVENTIONS:
Behavioral: Digital pre-therapy patient education program (StartHjelp) — After randomization the intervention group receives access to a pre-therapy informational app, presenting information about the treatment process, options, patient rights, user organizations, and self-help while on waiting list before mental health outpatient treatment. The information is presented stepwise through video and text, while also providing links to additional information if needed. The videos are made available to the patients gradually, with more general information about the treatment process first, and more specific information as the first session approaches. The patient has the opportunity to rewatch the videos as they please.
  Arms: Digital pre-therapy informational intervention (StartHjelp).
Behavioral: Comparator intervention — After randomization, while on waiting list, the control group gets sent all the same information as the intervention group in written form, by mail.
  Arms: Control group

SUMMARY:
Community mental health centers (CMHCs) face significant challenges in meeting the needs of individuals with mental health issues. For example, due to high demand, there are long waiting lists and low engagement rates. Innovative interventions are urgently needed to address these challenges to improve patient engagement, coping skills, and overall health outcomes. Educational and self-management interventions have shown promise in enhancing patient activation and treatment satisfaction in other contexts. They may therefore be potential solutions to reduce the identified challenges in the mental health service. To bridge these knowledge and practice gaps, this study aims to evaluate a digital pre-therapy patient education program tailored specifically for adults with mental disorders. This intervention aims to enhance treatment satisfaction, patient activation, knowledge, patient engagement, and overall mental health outcomes.

DETAILED DESCRIPTION:
Community mental health centers (CMHCs) play a pivotal role in the provision of comprehensive care and support for individuals with mental health challenges. However, these centers often face formidable obstacles, including surging patient demands, lengthy waiting lists, high dropout rates, and barriers to engagement, stigma, and negative attitudes. Given these challenges, there exists an urgent imperative to develop innovative interventions that can enhance treatment satisfaction, patient activation, knowledge, and patient engagement, and ultimately yield improved mental health outcomes. One promising approach for addressing these challenges lies in the realm of patient engagement and enablement strategies, particularly through the implementation of digital educational interventions.

The investigators hypothesize that utilizing innovative technology to deliver an early digital self-management educational program improves treatment satisfaction, patient activation, knowledge, patient engagement, and overall mental health outcomes without substantially increasing service costs. The impact of utilizing innovative technology to deliver an early digital pre-therapy patient education program through the HelsaMi web patient portal is promising. By leveraging technology, it is possible to reach a wider audience and provide accessible and convenient information, with the same standard to all patients. This approach has the potential to improve patient outcomes, increase treatment adherence, and reduce the burden on healthcare resources. By demonstrating the benefits of digital interventions, our research will pave the way for more efficient and cost-effective mental healthcare services, benefiting both patients and healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Put on the waiting list for mental health outpatient treatment in the active study period.
* Willing to participate in the study
* Over 18 years
* Understand written and spoken Norwegian

Exclusion Criteria:

* In need of acute help

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | measured on T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Patient satisfaction with the client satisfaction questionnaire (CSQ). The CSQ prompts the patient to evaluate different aspects of the care received with an 4 point ordinal scale (very dissatisfied, somewhat dissatisfied, somewhat satisfied, very satisfied).
Patient activation | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Patient activation measure 13 will be used. This questionaire measures patient activation by asking about knowledge, skills, and ability to manage one's own health, and health care usage. It consists of 13 items which is answered on an 4 point ordinal scale (Strongly disagree, somewhat disagree, somewhat agree, and strongly agree. Respondents have the option to answer "not applicable to me" as well.
Knowledge and treatment preferences | measured on T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks)
  Knowledge will be measured by five questions. All questions are introduced by "how much knowledge do you have about" (how outpatient clinics work; what happens in therapy; self management and user participation; patient rights; treatment options available to you). These questions are answered on a six-point ordinal scale ranging from "Nothing" to "Very much". After these 5 questions a follow up question "do you know what type of treatment you want?", answered either "yes", "no", or "don't know", is asked. If the answer is "yes" the patient is prompted to write what it is that they want.

SECONDARY OUTCOMES:
Patient enablement | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  To measure patient enablement the PEN-13 will be used. The PEN-13 is a 13 item questionnaire which measure patient enablement across two domains (patient practitioner interaction and self management). The answers are given on a five-point Likert scale (strongly disagree, disagree, neither/nor, agree, and strongly agree).
Level of functioning | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Work and social adjustment, or level of functioning, is measured by the Work and Social Adjustment Scale (WSAS). The WSAS have five items that measure functioning across different domains: Work, home management, social leisure activities, private leisure activities, and close relationships. Each question is answered on a 0 to 8 scale, where 0 means "not at all" impaired, and 8 means "very severely" impaired.
Mental health | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Mental health will be measured the Patient Health questionnaire 4. A four-item questionnaire with two items measuring the severity of anxiety symptoms and two items measuring the severity of depression symptoms.
Perceived stress | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Perceived stress will be measured by Perceived stress Scale-4, which comprise of four items scored on a five-point ordinal scale scored 0-4. Answers range from Never to very often.
Health related Quality of life | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Health related quality of life will be measured with the EQ-5D-5L. This questionnaire measure health related quality of life with five items, where each items prompts the patient to evaluate their "problem level" across a specific domain (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Question responses are ordinal and include "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". Respondents are also asked to rate their health on a 0-100 scale.
Intentions for patient involvement | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks), T2 (after intervention; up to 8 weeks), T3 (12 months follow up; up to 60 weeks)
  Intentions for patient involvement were measured by asking the question "How much do you want to participate in decisions related to your treatment measured on a six point ordinal scale ranging from "nothing" to "very much".
Expectations | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks)
  To investigate patients' expectations about the interventions an open question "What are your expectations for this intervention".

OTHER OUTCOMES:
Costs | T4 (24 months follow up; up to 112 weeks)
  Cost of app development and maintenance are being tracked to compare it against its outcomes to evaluate its cost-benefit.
App engagement | T2 (after intervention; up to 8 weeks)
  To measure app engagement, anonymized data of app usage will be gathered through the app itself.
health care usage | T4 (24 months follow up; up to 112 weeks)
  Data from official patient registries will be used to track (drop out, number of consultations, type of treatment)
System usability | T2 (after intervention; up to 8 weeks)
  To test the usability of the app itself the System Usability Scale will be used, a widely used 10-item scale that measure how the user experience using and trying to understand a digital tool.
Alcohol use disorder test | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks)
  To screen for alcohol use disorders Alcohol Use Disorders Identification Test (AUDIT) will be used. AUDIT has 10 items and uses the last 12 months as a reference for answering.
Drug use disorder test | measured on T0 (baseline; at 0 weeks), T1 (after randomization, before intervention; up to 2 weeks)
  To screen for drug use disorders Drug Use Disorders Identification Test (DUDIT) will be used. DUDIT has 11 items and uses the last 12 months as a reference for answering.
Work status | T4 (24 months follow up; up to 112 weeks)
  Data from official patient registries will be used to track work status (disability status, employment or sick leave).

CONTACTS AND LOCATIONS:
Overall Officials: Mariela L. Lara-Cabrera, Principal Investigator — St.Olavs Hospital and Norwegian University of Science and Technology (NTNU); Rolf W. Gråwe, PhD, Prof., Study Chair — St.Olavs Hospital and Norwegian University of Science and Technology (NTNU)
Locations (1):
- St.Olavs Hospital, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No